CLINICAL TRIAL: NCT03006718
Title: SCD-PROMIS: A Software Platform to Enhance Self-efficacy and Patient-provider Engagement for Patients With Sickle Cell Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julia Finkel (Other)
Collaborators: Arizona State University (Other); Children's National Research Institute (Other)
Responsible Party: Sponsor-Investigator, Julia Finkel, ANESTHESIOLOGIST, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7618
Record Dates: First submitted 2016-12-22; First posted 2016-12-30 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Sickle Cell Disease; Anemia; Anemia, Hemolytic; Anemia, Sickle Cell; Hematologic Diseases
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia; Anemia, Hemolytic; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental): Participants must have SCD (HbSS, HbSC, HbSβ0 thalassemia, HbSβ+ thalassemia, HbSOArab), within the age range of 8 - 21 years, and be admitted to the hospital for vaso-occlusive crisis (VOE)-related pain. The investigators will also collect Proxy PROMIS measures from parents of participants between the ages of 8 and 17-years who have agreed to participate in the study.
  All participants will use the PROMIS for Pain Management App over 5 consecutive weeks (starting at hospital discharge).
  Interventions: Other: PROMIS for Pain Management App

INTERVENTIONS:
Other: PROMIS for Pain Management App — At hospital discharge, the investigators will collect baseline surveys, a blood sample, and download the PROMIS for Pain Management App onto the subject's mobile device. For five consecutive weeks, PROMIS measures will be collected through weekly surveys. The investigators plan to compensate patients for their time. Patients will come back to the hospital after 35 days for a final blood draw and set of surveys. In the event a patient gets readmitted, the investigators will record that admission. The investigators will also collect Proxy PROMIS measures from parents of participants between the ages of 8 and 17-years who have agreed to participate in the study. It is the goal of the investigators to engage one of the parents in the reporting of weekly validated Proxy PROMIS measures.
  Other Names: SCD-PROMIS

SUMMARY:
The overall goal of the project is to reduce pain-related, 30-day readmission rates for sickle cell disease (SCD) patients. The investigators want to see if a mobile phone application (app) can help decrease the need for repeat admission to the hospital because of sickle cell pain.

DETAILED DESCRIPTION:
Pain is the main reason why SCD patients are admitted and readmitted to the hospital. In fact, readmission rates of SCD patients are higher than those of asthmatics and diabetics. In order to reduce 30-day hospital readmission rates and improve patient care quality, the Affordable Care Act and Centers for Medicare and Medicaid Services have established the Readmissions Reduction Program. In keeping with this effort, the investigators propose a methodology and supporting technology that has the potential to change the way SCD patients are monitored after hospital discharge and in turn, decrease readmission rates. This methodology also has the potential to enhance the quality of life of SCD patients by improving patient reporting, self-efficacy, and increasing patient/provider engagement when there is worsening pain and increased admission/readmission risk. This software platform uses validated Patient Reported Outcome Measurement Information System (PROMIS) measures to remotely monitor SCD patients' pain and related outcomes after hospital discharge. With this initial study, the investigators propose to use this monitoring platform to identify the predictors of readmission, to develop a readmission prediction engine, and to design the next version of the app with built in interventions to address those readmission risks. This monitoring platform could also increase healthcare provider engagement when there is a worsening of patients' pain and/or an increased risk of readmission. In order to build and optimize this monitoring platform, the investigators have assembled a team of engineers, hematologists, pain researchers, and statisticians that have worked together, and who collectively have the expertise to develop and test the feasibility and predictive value of the application in a large population of SCD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with Sickle Cell Disease (SCD) (HbSS, HbSC, HbSβ0 thalassemia, HbSβ+ thalassemia, HbSOArab) admitted to the hospital for vaso-occlusive crisis (VOE)-related pain within the age range of 8 - 21 years.
2. Ability to provide informed consent/assent, comply with study related procedures, evaluations, and follow-up. In the event that a patient does not have a smart mobile device (i.e., one that can support the study application), one will be provided for the patient. Patients younger than the age of 11 years may use their parents phone if they do not have one. If a patient has a smart mobile device but their parent does not want them to use the device for the study, the patient may use their parent's phone instead.
3. Parent of participants with SCD (HbSS, HbSC, HbSβ0 thalassemia, HbSβ+ thalassemia HbSOArab) admitted to the hospital for vaso-occlusive crisis (VOE)-related pain within the age range of 8 - 17 years who has assented to participate in the study.
4. Ability to provide informed consent, comply with study related procedures, evaluations, and follow-up. In the event that a parent does not have a mobile device, one will be provided for the duration of the study.

Exclusion Criteria:

1. Inability to give informed consent/assent as determined by the investigators
2. Patients with SCD who were admitted for reasons other than VOE-related pain
3. Parents of patients with SCD who were admitted for reasons other than VOE-related pain or do not assent to participate

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Readmission rate | 35 days
  The investigators want to determine if the use of this mobile app by itself reduces readmission rates. The investigators will compare the readmission rate of patients who use this mobile app with those who do not.
Readmission risk | 35 days
  The rate of hospital readmission will be estimated by time periods (e.g., 1, 2, 3, and 4 weeks after discharge).

SECONDARY OUTCOMES:
Patient Compliance | 35 days
  To evaluate our app design features, the investigators will track each user's interaction with the app for post-analysis to determine time spent answering the questions and the value of reminders. It is the investigators intent to determine if features will be used as intended by the app design.
Patient Usability | 35 days
  At the end of five weeks the investigators will administer a survey to parents and participants to determine the usability of this app.This information will lead to improvements on the design of future iterations of the app.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Finkel, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No